CLINICAL TRIAL: NCT00301379
Title: Prospective Registry Study of Neoadjuvant Therapy in Conjunction With Liver Transplantation for Cholangiocarcinoma
Brief Title: Registry Study of Neoadjuvant Chemoradiation & Transplant for Cholangiocarcinoma Patients
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 05-0651 / 201102096
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Observational
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with unresectable cholangiocarcinoma.
  Interventions: Other: Observation data collection study.

INTERVENTIONS:
Other: Observation data collection study. — This is a data collection study where the main purpose is to collect information about the treatments patients receive for their unresectable cholangiocarcinoma.

SUMMARY:
This is an observational study intended to validate results of a previous study done at the Mayo Clinic. Patients are treated with combination chemotherapy and radiation and maintained on oral Xeloda until they can receive liver transplant. A staging laparotomy is performed before chemoradiation in order to identify patients who will most benefit from the treatment and to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cholangiocarcinoma that has been established preoperatively by at least one of the following criteria:

   1. A positive brush cytology or biopsy result obtained at the time of cholangiography;
   2. Fluorescence in situ hybridization demonstrating aneuploidy;
   3. A serum CA 19-9 value greater than 100 U/mL in the presence of a radiographically characteristic malignant stricture in the absence of cholangitis.
   4. Listed for OLT for hilar cholangiocarcinoma
2. Tumor/stricture is above the cystic duct and is unresectable.
3. A suitable candidate for orthotopic liver transplantation as judged by the liver transplant team. All 3 treatment modalities are not needed to confirm eligibility for this registry trial.
4. >/= 18 years of age.
5. Willing and able to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2005-08-12 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients withdrawn due to toxicity and other treatment related events. | Completion of treatment for all patients (estimated to be 18 years total)

SECONDARY OUTCOMES:
Proportion of patients who respond to treatment | Completion of treatment for all patients (estimated to be 18 years total)
  -Response is defined as an absence of progressive disease or metastasis, so that the patient remains a candidate for liver transplantation
Overall survival | Completion of treatment for all patients (estimated to be 18 years total)
Disease-free survival | Completion of treatment for all patients (estimated to be 18 years total)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Chapman, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heimbach JK, Haddock MG, Alberts SR, Nyberg SL, Ishitani MB, Rosen CB, Gores GJ. Transplantation for hilar cholangiocarcinoma. Liver Transpl. 2004 Oct;10(10 Suppl 2):S65-8. doi: 10.1002/lt.20266. PMID 15382214
- [Background] Jarnagin WR, Fong Y, DeMatteo RP, Gonen M, Burke EC, Bodniewicz BS J, Youssef BA M, Klimstra D, Blumgart LH. Staging, resectability, and outcome in 225 patients with hilar cholangiocarcinoma. Ann Surg. 2001 Oct;234(4):507-17; discussion 517-9. doi: 10.1097/00000658-200110000-00010. PMID 11573044
- [Background] Casavilla FA, Marsh JW, Iwatsuki S, Todo S, Lee RG, Madariaga JR, Pinna A, Dvorchik I, Fung JJ, Starzl TE. Hepatic resection and transplantation for peripheral cholangiocarcinoma. J Am Coll Surg. 1997 Nov;185(5):429-36. doi: 10.1016/s1072-7515(97)00088-4. PMID 9358085
- [Background] De Vreede I, Steers JL, Burch PA, Rosen CB, Gunderson LL, Haddock MG, Burgart L, Gores GJ. Prolonged disease-free survival after orthotopic liver transplantation plus adjuvant chemoirradiation for cholangiocarcinoma. Liver Transpl. 2000 May;6(3):309-16. doi: 10.1053/lv.2000.6143. PMID 10827231
- [Background] Brandsaeter B, Isoniemi H, Broome U, Olausson M, Backman L, Hansen B, Schrumpf E, Oksanen A, Ericzon BG, Hockerstedt K, Makisalo H, Kirkegaard P, Friman S, Bjoro K. Liver transplantation for primary sclerosing cholangitis; predictors and consequences of hepatobiliary malignancy. J Hepatol. 2004 May;40(5):815-22. doi: 10.1016/j.jhep.2004.01.002. PMID 15094230
- [Background] Madariaga JR, Iwatsuki S, Todo S, Lee RG, Irish W, Starzl TE. Liver resection for hilar and peripheral cholangiocarcinomas: a study of 62 cases. Ann Surg. 1998 Jan;227(1):70-9. doi: 10.1097/00000658-199801000-00011. PMID 9445113
- [Background] Shimoda M, Farmer DG, Colquhoun SD, Rosove M, Ghobrial RM, Yersiz H, Chen P, Busuttil RW. Liver transplantation for cholangiocellular carcinoma: analysis of a single-center experience and review of the literature. Liver Transpl. 2001 Dec;7(12):1023-33. doi: 10.1053/jlts.2001.29419. PMID 11753904
- [Background] Goldstein RM, Stone M, Tillery GW, Senzer N, Levy M, Husberg BS, Gonwa T, Klintmalm G. Is liver transplantation indicated for cholangiocarcinoma? Am J Surg. 1993 Dec;166(6):768-71; discussion 771-2. doi: 10.1016/s0002-9610(05)80696-8. PMID 8273866
- [Background] Hassoun Z, Gores GJ, Rosen CB. Preliminary experience with liver transplantation in selected patients with unresectable hilar cholangiocarcinoma. Surg Oncol Clin N Am. 2002 Oct;11(4):909-21. doi: 10.1016/s1055-3207(02)00036-4. PMID 12607579
- [Background] Sudan D, DeRoover A, Chinnakotla S, Fox I, Shaw B Jr, McCashland T, Sorrell M, Tempero M, Langnas A. Radiochemotherapy and transplantation allow long-term survival for nonresectable hilar cholangiocarcinoma. Am J Transplant. 2002 Sep;2(8):774-9. doi: 10.1034/j.1600-6143.2002.20812.x. PMID 12243499
- [Background] Tsavaris, Inv New Drugs, 22:193, 2004;Verdarame, Anti-Cancer Drugs, 11:707,2000.
- [Background] Picus, Proc ASCO, 13:208, 1994.
- [Background] Broome U, Olsson R, Loof L, Bodemar G, Hultcrantz R, Danielsson A, Prytz H, Sandberg-Gertzen H, Wallerstedt S, Lindberg G. Natural history and prognostic factors in 305 Swedish patients with primary sclerosing cholangitis. Gut. 1996 Apr;38(4):610-5. doi: 10.1136/gut.38.4.610. PMID 8707097
- [Background] Valle JW WH, Palmer DD, Cunningham D, Anthoney DA, Maraveyas A, Hughes SK, Roughton JA, Bridgewater JA: Gemcitabine with or without cisplatin in patients (pts) with advanced or metastatic biliary tract cancer (ABC): Results of a multicenter, randomized phase III trial (the UK ABC-02 trial). J Clin Oncol 27:15s, 2009 (suppl, abstr 4503), 2009
- [Background] Williams KJ, Picus J, Trinkhaus K, Fournier CC, Suresh R, James JS, Tan BR. Gemcitabine with carboplatin for advanced biliary tract cancers: a phase II single institution study. HPB (Oxford). 2010 Aug;12(6):418-26. doi: 10.1111/j.1477-2574.2010.00197.x. PMID 20662793
- [Background] Harder J, Riecken B, Kummer O, Lohrmann C, Otto F, Usadel H, Geissler M, Opitz O, Henss H. Outpatient chemotherapy with gemcitabine and oxaliplatin in patients with biliary tract cancer. Br J Cancer. 2006 Oct 9;95(7):848-52. doi: 10.1038/sj.bjc.6603334. Epub 2006 Sep 12. PMID 16969352
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu